CLINICAL TRIAL: NCT01081704
Title: A Study to Evaluate the Pharmacokinetics of Ustekinumab Following a Single Subcutaneous Administration of 45 mg or 90 mg to Healthy, Chinese, Male Subjects
Brief Title: A Study of the Pharmacokinetics of Ustekinumab in Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016207
Record Dates: First submitted 2010-02-25; First posted 2010-03-05 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Healthy volunteer; Chinese male; Stelara
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): ustekinumab Single dose of 45 mg subcutaneous injection
  Interventions: Drug: ustekinumab
- 002 (Experimental): ustekinumab Single dose of 90 mg subcutaneous injection
  Interventions: Drug: ustekinumab

INTERVENTIONS:
Drug: ustekinumab — Single dose of 45 mg subcutaneous injection
  Arms: 001
Drug: ustekinumab — Single dose of 90 mg subcutaneous injection
  Arms: 002

SUMMARY:
A study of the pharmacokinetics of ustekinumab in Chinese male subjects.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned by chance), open-label (both the physician and subject know the assigned study medication) study to assess the safety, tolerability, immune response, pharmacokinetics (what the body does to the drug), of ustekinumab (Stelara). The study population will consist of 24 healthy male participants in China. Participants will receive a single dose of either 45mg or 90 mg ustekinumab. Participants will be in the study for up to 16 weeks. Safety assessments will be performed throughout the study and include obtaining and evaluating laboratory tests, vital signs (e.g., blood pressure), and the occurrence and severity of adverse events. A single dose of 45 mg or 90 mg ustekinumab.

ELIGIBILITY:
Inclusion Criteria:

* Have no clinically relevant abnormalities
* Non smoker

Exclusion Criteria:

* Have or had a history of clinically significant, severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease
* Have any underlying physical or psychological medical condition
* Be unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access to veins

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Determine what the body does to ustekinumab (pharmacokinetics) in Chinese Male participants. | Week 16

SECONDARY OUTCOMES:
Safety and tolerability of ustekinumab by evaluating laboratory tests, vital signs (e.g., blood pressure), and the occurrence and severity of adverse events | Week 16
Immune response (immunogenicity) of ustekinumab | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (1):
- Beijing, China

REFERENCES:
- [Derived] Zhu Y, Wang Q, Frederick B, Bouman-Thio E, Marini JC, Keen M, Petty KJ, Davis HM, Zhou H. Comparison of the pharmacokinetics of subcutaneous ustekinumab between Chinese and non-Chinese healthy male subjects across two Phase 1 studies. Clin Drug Investig. 2013 Apr;33(4):291-301. doi: 10.1007/s40261-013-0072-2. PMID 23512638